CLINICAL TRIAL: NCT06730932
Title: A Prospective，Single Arm, Multicenter Clinical Study of BTLA Monoclonal Antibody JS004 (B/T Lymphocyte Attenuator Factor Monoclonal Antibody) in Combination With Toripalimab in Patients With Unresectable or Advanced Renal Cell Carcinoma Who Had Failed Previous Immunotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCC-IIT-JS004-S01
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Unresectable or Advanced Clear Cell Renal Cell Carcinoma That Has Progressed After Previous Immunotherapy
Keywords: JS004; Toripalimab; ccRCC; immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS004 combine with Toripalimab (Experimental)
  Interventions: Drug: JS004（BTLA monoclonal antibody，intravenously）,Toripalimab（ anti-PD-1specific antibody，intravenously)

INTERVENTIONS:
Drug: JS004（BTLA monoclonal antibody，intravenously）,Toripalimab（ anti-PD-1specific antibody，intravenously) — Recombinant humanized anti-BTLA monoclonal antibody (JS004) injection 200mg via IV infusion once every 3 weeks
  Toripalimab 240mg via IV infusion once every 3 weeks
  JS004 will be administered in combination with toripalimab until disease progression or intolerable toxicity or up to 2 years of treatment or other reasons specified in the protocol

SUMMARY:
This study is A prospective，single arm, multicenter clinical study of BTLA monoclonal antibody JS004 (B/T lymphocyte attenuator factor monoclonal antibody) in combination with toripalimab in patients with unresectable or advanced renal cell carcinoma who had failed previous immunotherapy Subjects will receive JS004（B/T lymphocyte attenuator factor monoclonal antibody） plus Toripalimab until disease progression, development of unacceptable toxic effects, death, a decision by the physician or patient to withdraw from the trial. The primary endpoint is ORR per RECIST v1.1 as assessed by investigators(continuous treatment for up to 2 years).

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood and voluntarily signed the Informed Consent Form (ICF);
2. 18-75 years old (at the time of signing the informed consent form); No gender restrictions; ECOG PS score: 0-1 points;
3. Renal cell carcinoma with clear cell components confirmed by histology or cell pathology, including metastatic renal cell carcinoma mainly composed of clear cell components;
4. Previous treatment history of the subject: Patients who have received 1-2 systemic treatments containing immunotherapy and have experienced disease progression or intolerance;
5. Confirm the presence of at least one measurable lesion according to RECIST 1.1 criteria;
6. Agree to provide sufficient previously stored tumor tissue specimens or agree to undergo biopsy

Collect tumor tissue for PD-L1, CD8 expression level determination, and MSI, TMB, KRAS, BRAF, PIK3CA, NRAS, PTEN, EGFR, HER2, HRAS, KIT, MET, ROS1, POLE, POLD1, TP53 gene mutation detection; 7. The main organ functions well and meets the following standards:

1. Blood routine examination standards (corrected for no blood transfusion or use of hematopoietic stimulating factor drugs within 2 weeks before the first trial medication):

   1. Hemoglobin (HGB) ≥ 90g/L;
   2. Absolute neutrophil count (NEUT) ≥ 1.5 × 109/L;
   3. Platelet count (PLT) ≥ 100 × 109/L.
2. Biochemical tests must meet the following standards:

   1. Serum total bilirubin (TBIL) ≤ 1.5 × ULN or direct bilirubin ≤ 1.0 × ULN;
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN. If accompanied by liver metastasis, ALT and AST should be ≤ 5 × ULN;
   3. Serum creatinine (CR) ≤ 1.5 × ULN or creatinine clearance rate (CCR) ≥ 60ml/min
3. Coagulation function test:

   Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN, unless the subject is receiving anticoagulant therapy and coagulation parameters (PT/INR and APTT) are within the expected range of anticoagulant therapy at screening;
4. Left ventricular ejection fraction (LVEF) ≥ 50%;
5. Endocrine function: Normal thyroid stimulating hormone (TSH), or abnormal TSH but normal FT3 and FT4; 8. Willing and able to comply with the research plan's visits, treatment laboratory tests, sample collection, and other procedures; 9. Female patients with fertility must voluntarily adopt efficient contraceptive measures (such as oral contraception, injection contraception, or implanted barrier contraception, spermicides and condoms, or intrauterine devices) for at least 120 days from the last dose during the study period, and have negative urine or serum pregnancy test results ≤ 7 days before enrollment; 10. Male patients who have not been sterilized must voluntarily adopt effective contraceptive measures for at least 120 days from the last dose during the study period.

Exclusion Criteria:

Participants who meet any of the following criteria will not be allowed to enter this study:

1. History of malignant tumors other than the research disease within the past 5 years, except for malignant tumors that can be expected to recover after treatment (including but not limited to fully treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell carcinoma, or radical surgery for ductal carcinoma in situ);
2. Four weeks before the first study medication, receive systemic treatment with other anti-tumor drugs (if it has a half-life of five, it can be included in the group), or receive local anti-tumor treatment, or receive clinical investigational drug or device treatment;
3. Received immunotherapy within 4 weeks prior to the first study medication;
4. Have undergone major surgery (as determined by the investigator) or are in the recovery period within 4 weeks prior to the first trial administration;
5. Patients who have previously received treatment with anti BTLA or anti HVEM antibodies;
6. Have a history of severe drug allergies, including but not limited to antibody drugs;
7. Patients with contraindications for immunotherapy restart: a) grade 2-4 immune myocarditis; b) Severe grade 4 proteinuria; c) Severe or life-threatening grade 4 immune hepatitis; d) Severe grade 3-4 immune pneumonia; e) Severe inflammatory arthritis that significantly affects daily life or quality of life; f) Severe neurological toxicity: grade 2-4 myasthenia gravis; Any level of Guillain Barr é syndrome (GBS) or transverse myelitis; Grade 2-4 encephalitis; g) Severe or life-threatening grade 3-4 pancreatitis; h) Serious or life-threatening bullous diseases (grades 3-4); i) Severe grade 3-4 uveitis or episcleritis;
8. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation, or requiring long-term treatment with corticosteroids;
9. Only hypothyroidism, suprarenal or pituitary dysfunction that can be controlled by hormone replacement therapy, type I diabetes, psoriasis or vitiligo that does not need systematic treatment can participate in this study;
10. The toxicity has not improved after previous anti-tumor treatment, that is, it has regressed to baseline, NCI-CTCAE 5.0 grade 0-1 (except for hair loss), or the level specified in the inclusion/exclusion criteria. Irreversible toxicity (such as hearing loss) that is reasonably expected not to be exacerbated by the investigational drug can be included in this study;
11. Suffering from central nervous system metastasis and/or malignant meningitis. Subjects who have received treatment for brain metastases may be considered for participation in this study, provided that their condition has been stable for at least 3 months, no disease progression has been confirmed by imaging examinations within 4 weeks prior to the first administration of the study, all neurological symptoms have returned to baseline levels, there is no evidence of new or expanded brain metastases, and radiation, surgery, or steroid therapy has been discontinued at least 28 days prior to the first administration of the study treatment;
12. The known history of liver diseases with clinical significance, including those with active viral hepatitis (when hepatitis B virus surface antigen (HBsAg) and or hepatitis B virus core antibody (HbcAb) are positive, hepatitis B B virus (HBV) DNA>10000 copies/mL or>2000 IU/mL; Hepatitis C virus (HCV) antibody positive and HCV RNA positive, or other active hepatitis, clinically significant moderate to severe cirrhosis;
13. Patients with uncontrolled third interstitial fluid accumulation that requires repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (patients who do not require drainage or have no significant increase in fluid accumulation after stopping drainage for 3 days can be enrolled);
14. Corticosteroid drugs (prednisone>10mg/day or equivalent dose) or other immunosuppressive drugs received systemically within 14 days prior to the first study medication;
15. Patients with any severe and/or uncontrolled illnesses, including:

    1. Hypertension that cannot be well controlled with antihypertensive medication (systolic blood pressure>140 mmHg or diastolic blood pressure>90 mmHg);
    2. Unstable angina or myocardial infarction, coronary artery bypass grafting or stent implantation within 6 months prior to study medication;
    3. Suffering from grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480ms), and grade ≥ 2 congestive heart failure (NYHA classification); Grade II or above heart conduction block; Left ventricular ejection fraction (LVEF)<50%;
    4. Poor control of diabetes (FBG>10 mmol/L);
    5. Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0g;
    6. Active or uncontrolled severe infections;
16. Suffering from or suspected to have active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc;
17. Renal failure requires hemodialysis or peritoneal dialysis;
18. Individuals with a history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
19. History of receiving attenuated live vaccines within 4 weeks prior to the first study medication or expected to receive attenuated live vaccines during the study period;
20. Individuals with a history of substance abuse and inability to quit, or those with a history of mental disorders;
21. Pregnant or lactating women;
22. Based on the researcher's assessment, there may be other severe, acute, or chronic medical or mental illnesses or laboratory abnormalities that could increase the risk of participating in the study or interfere with the interpretation of the research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR per RECIST v1.1 as assessed by investigators | Up to 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Disease control rate (DCR) | Up to 2 years
  Disease control rate (DCR) assessed according to RECIST v1.1
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment until death due to any cause.

OTHER OUTCOMES:
Adverse Event | Up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0, also types and degree

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No